CLINICAL TRIAL: NCT07085806
Title: Effect of Pentoxifylline on Liver Regeneration After Right Lobe Donor Hepatectomy: A Randomized Control Trial
Brief Title: To Study Effect of Injection Pentoxifylline on Liver Growth After Major Liver Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IEC/2024/110/MA01
Record Dates: First submitted 2025-05-29; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-05

CONDITIONS: Liver Regeneration
Keywords: Role of Injection pentoxifylline in Liver regeneration after Right lobe Hepatectomy
MeSH Terms: interventions — Pentoxifylline; Plasmalyte A

STUDY DESIGN:
Intervention Model Description: Randomised Control Trial- open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasmalyte (Active Comparator): Intravenous fluid plasmalyte.
  Interventions: Other: Plasmalyte
- Pentoxifylline group (Experimental): Intravenous injection Pentoxifylline
  Interventions: Drug: Pentoxifylline (also known as oxpentifylline)

INTERVENTIONS:
Drug: Pentoxifylline (also known as oxpentifylline) — Intravenous injection Pentoxifylline 1 mg/kg/hr dissolved in Plasma Lyte/0.9% Normal saline from12 hours before the surgery to 72 hours after the Surgery
  Arms: Pentoxifylline group
Other: Plasmalyte — Plasmalyte
  Arms: Plasmalyte

SUMMARY:
Posthepatectomy liver failure (PHLF) remains a significant life-threatening problem after major hepatectomies. Pentoxifylline is shown to have potent vasodilating properties for peripheral blood vessels, along with the hepatic vasculature. In a Double-blinded, randomized, controlled trial (RCT) at a single tertiary care center (2006-2009) by Petrowsky, Henrik et al (Annals of Surgery, November 2010) on 101 Non-cirrhotic patients undergoing major Hepatectomy, they demonstrated beneficial effects of Pentoxifylline on regeneration of small remnant livers (RLBW ratio ≤ 1.2%). In mice model, pentoxifylline (Tian, Yinghua, et al Proceedings of the National Academy of Sciences 103.12 (2006)) is shown to confer protective effects against small-for-size syndrome in arterialized small-for-size liver transplantation. This Randomised control trial is being conducted to analyze the effect of Pentoxifylline supplementation in live donors undergoing donor hepatectomy with respect to markers of anatomical regeneration in a high volume liver transplant center in India.

ELIGIBILITY:
Inclusion Criteria:

* All live donors undergoing Right Donor Hepatectomy after ethical board clearance in the Department of HPB Surgery and Liver Transplantation

Exclusion Criteria:

* Negative consent Hypersensitivity to Pentoxifylline

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
To assess effect of Pentoxifylline supplementation on Anatomical (Volume) Regeneration of liver in the Perioperative period (POD-14) in Right lobe donor Hepatectomy | 2 weeks post-operatively
  Regenerated liver volume post-surgery Day-14 and Percentage of volume restored after Post surgery day 14 as compared to pre-operatively calculated Remnaant liver volume

SECONDARY OUTCOMES:
To evaluate the effect of Pentoxifylline on Serum Bilirubin- Time to Normalization | 2 weeks
  Serum bilirubin on Post-operative Day 1 to 7 and 14
To evaluate the effect on HGF | 1 week
  HGF (Hepatocyte Growth Factor) levels on Baseline, Postoperative Day 3, and Day 7
To study the effect of Pentoxifylline supplementation on post-operative complications in donor right hepatectomy | Postoperative Day 14
  Clavien-Dindo Classification Grading on Post-operative Day 14
Time to normalziation of Aspartate Transaminase | Post-operative Day 14
  Aspartate transaminase (Baseline, Post-operative Day 1 to 7 and 14)
Time to normalzation of Alanine transaminase | Post-operative Day 14
  Alanine Transaminase on BASELINE, POST-OPERATIVE DAY 1 TO 7 and 14
Time to Normalisation of International Normalized Ratio | Post-operative Day 14
  International Normalized Ratio on Baseline Post-operative Day 1 to 7 and 14
Time to normalisation of Serum Alkaline phosphatase | Post-operative Day 14
  Serum Alkaline Phosphatase levels on Baseline, Post-operative Day 1 to 7 and 14
Time to normalisation of Gamma-Glutamyl Transferase | Post-operative Day 14
  Gamma-Glutamyl Transferase levels on baseline, Post-operative Day 1 to 7 and 14
Effect on TNF-alpha (Tumor Necrosis Factor alpha) | Post-operative Day 7
  TNF-alpha (Tumor Necrosis Factor alpha) levels on Baseline, Post-operative Day 3 and 7
Effect on IL-6 (Interleukin-6) | Post-operative day 7
  IL-6 levels on baseline , post-operative day 3 and 7
Effect on TGF-beta (Transforming Growth Factor beta) | POst-operative Day 7
  TGF-beta levels on Baseline, Post-operative Day 3 and 7
Effect on AFP (Alpha-fetoprotein) | Post-operative day 7
  AFP (Alpha-fetoprotein) levels on Baseline, post-operative Day 3 and Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tian Y, Jochum W, Georgiev P, Moritz W, Graf R, Clavien PA. Kupffer cell-dependent TNF-alpha signaling mediates injury in the arterialized small-for-size liver transplantation in the mouse. Proc Natl Acad Sci U S A. 2006 Mar 21;103(12):4598-603. doi: 10.1073/pnas.0600499103. Epub 2006 Mar 13. PMID 16537374
- [Result] Martino RB, Coelho AM, Kubrusly MS, Leitao R, Sampietre SN, Machado MC, Bacchella T, D'Albuquerque LA. Pentoxifylline improves liver regeneration through down-regulation of TNF-alpha synthesis and TGF-beta1 gene expression. World J Gastrointest Surg. 2012 Jun 27;4(6):146-51. doi: 10.4240/wjgs.v4.i6.146. PMID 22816029
- [Result] Petrowsky H, Breitenstein S, Slankamenac K, Vetter D, Lehmann K, Heinrich S, DeOliveira ML, Jochum W, Weishaupt D, Frauenfelder T, Graf R, Clavien PA. Effects of pentoxifylline on liver regeneration: a double-blinded, randomized, controlled trial in 101 patients undergoing major liver resection. Ann Surg. 2010 Nov;252(5):813-22. doi: 10.1097/SLA.0b013e3181fcbc5e. PMID 21037437